CLINICAL TRIAL: NCT05598502
Title: A Phase III, Open-label, Randomized Clinical Trial to Evaluate Efficacy and Safety of Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in Life-threatening Postpartum Hemorrhage in Reducing Adverse Maternal Outcome in Uganda
Brief Title: REBOA in Life-threatening Postpartum Hemorrhage (PPH) in Uganda
Acronym: REBOA-PPH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: Makerere University (Other); Kawempe National Referral Hospital (Unknown); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); University of Liverpool (Other); University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mak-UiB 102
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Post-partum Hemorrhage
Keywords: REBOA; Resuscitative Endovascular Occlusion of the Aorta
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Individual randomization
Masking Description: The study statistician will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REBOA (Experimental): Addition of REBOA (Resuscitative Endovascular Occlusion of the Aorta)
  Interventions: Device: REBOA, Resuscitative Endovascular Occlusion of the Aorta; Other: National guidelines
- National guidelines (Active Comparator): Treatment according to Uganda national guidelines for post-partum hemorrhage.
  Interventions: Other: National guidelines

INTERVENTIONS:
Device: REBOA, Resuscitative Endovascular Occlusion of the Aorta — The balloon catheter is inserted via the common femoral artery in the groin, accessed under ultrasound guidance due to weak femoral pulses, and the puncture is done by the Seldinger technique. The balloon is inserted along a guidewire 25-30 cm, safely below the renal arteries, to be in the right place to stop pelvic hemorrhage including life-threatening post-partum hemorrhage
  Arms: REBOA
Other: National guidelines — Standard management of postpartum hemorrhage according to Uganda national guidelines

SUMMARY:
Background Maternal mortality rates in many low-income countries (LMICs) remain high. The most prominent cause is bleeding after birth, called postpartum haemorrhage (PPH). In a recent report from Uganda, bleeding is the cause of 42% of all maternal deaths in Uganda.

Large parts of the monitoring of mothers during active management of third stage of labour is aiming to prevent and early detect PPH and take relevant actions. In spite of this and sometimes in referring mothers to tertiary hospitals, mothers will end up in a challenging condition where quick action is needed. A new method has proven successful for such instances, the Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA). This is a procedure commonly used for trauma of the lower part of the body but rarely used for PPH. A balloon catheter is inserted via the femoral artery in the groin into the aorta and then being inflated. This will prevent blood from passing to the lower part of the body, including the uterus. It will stop the bleeding and allow for the obstetrician to take relevant action. This is a safe procedure for up to 1 hour of balloon occlusion time including repeated short balloon deflations.

Objective To assess the efficacy and safety of Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in life-threatening postpartum haemorrhage (PPH) in reducing adverse maternal outcome compared to standard of care in Uganda.

Study design, setting and population A phase IIb/III, open label, 1:1 randomized clinical trial will be conducted at Kawempe National Referral Hospital, Kampala, Uganda, to evaluate the efficacy and safety of Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in life-threatening postpartum haemorrhage (PPH) in reducing adverse maternal outcome compared to standard of care. The inclusion criteria are: a) women with life-threatening PPH and a systolic blood pressure equal to or less than 80 mmHg, b) written consent. The exclusion criterion is prior cardiac arrest or intra-abdominal pregnancy. The sample size of the trial will be 212 participants. Enrolment will follow a group sequential design approach with two interim analyses at 50% and 85% of the total sample size, and a final analysis with full sample size.

Utility of the study It is crucial to explore alternative modalities that could prevent adverse maternal outcomes in life-threatening postpartum haemorrhage in Uganda and the rest of the world.

DETAILED DESCRIPTION:
Background

Maternal mortality rates in many low-income countries (LMICs) remain high. The most prominent cause is bleeding after birth, called postpartum hemorrhage (PPH). In a recent report from Uganda, bleeding is the cause of 42% of all maternal deaths in Uganda.

Large parts of the monitoring of mothers during active management of third stage of labor is aiming to prevent and early detect PPH and take relevant actions. In spite of this and sometimes in referring mothers to tertiary hospitals, mothers will end up in a challenging condition where quick action is needed. A new method has proven successful for such instances, the Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA). This is a procedure commonly used for trauma of the lower part of the body but rarely used for PPH. In this trial, it is done by an anesthesiologist where a balloon catheter is inserted via the femoral artery in the groin into the aorta and then being inflated. This will prevent blood from passing to the lower part of the body, including the uterus. It will stop the bleeding and allow for the obstetrician to take relevant action. This is a safe procedure for up to 1 hour of inflation.

Objective

To assess the efficacy and safety of the use of Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in life-threatening postpartum hemorrhage (PPH) in reducing adverse maternal outcome compared to standard of care in Uganda.

Primary objectives

* To assess if the proportion of participants with either maternal death and/or emergency hysterectomy, can be decreased from 50 % in the comparator arm (using standard of care alone) to 30 % or less in the intervention arm (using standard of care plus REBOA).
* To assess the safety of REBOA in a national referral hospital in a low-income country like Uganda.

Secondary objectives

* To assess if the proportion of participants with either maternal death and/or emergency hysterectomy is lower in the intervention arm when excluding 'inevitable' hysterectomies due to either an irreparable uterine rupture, a pathological placenta growing into the uterus (placenta accreta, increta or percreta) or a pathological uterus, such as a bicorne uterus or one with very large fibroids.
* To assess if the proportion of participants with maternal deaths is lower in the intervention arm compared to the comparator arm.
* To assess if the proportion of participants with emergency hysterectomy, is lower in the intervention arm compared to the comparator arm.
* To assess if the number of participants with acute kidney injury 35is lower in the intervention arm compared to the comparator arm
* To assess if the number of blood transfusion units is lower in the intervention arm compared to the comparator arm.
* To assess if post-partum haemoglobin concentration is higher in in the intervention arm compared to the comparator arm.
* To assess the time to insert the REBOA.

Study design, setting and population The trial design will be a seamless phase IIb/III study. The study will start with a phase IIb study where the focus is on assessing the safety of REBOA use in a national referral hospital in a low-income country like Uganda. In this phase there will be 10 participants recruited consecutively to intervention arm (REBOA) without randomisation. The aim of the pilot phase is to demonstrate that the REBOA procedure is safe and feasible in the patient cohort.

The phase III trial is a randomised, controlled, open-label, superiority trial among women with life-threatening post-partum haemorrhage with two parallel arms and a primary endpoint of either death or hysterectomy. Individual randomisation will be performed as block randomization with a 1:1 allocation.

The trial will be conducted at Kawempe National Referral Hospital, Kampala, Uganda.

The sample size of the trial will be 212 participants. Enrolment will follow a group sequential design approach with two interim analyses at 1/2 and 85% of the total sample size, and a final analysis with full sample size.

Results from Norway indicate that REBOA could be an efficient way to prevent post-partum hemorrhage ending in an adverse outcome such as death or emergency hysterectomy. It is not clear whether these results can be reproduced in a low-income setting where PPH is more prevalent, and resources are scarce. The REBOA device could reduce the risk of adverse outcome such as death or emergency hysterectomy. It will be compared to standard of care.

Utility of the study

It is crucial to explore alternative modalities that could prevent adverse maternal outcomes in life-threatening postpartum hemorrhage in Uganda and the rest of the world.

ELIGIBILITY:
Inclusion Criteria:

* Patients with life-threatening PPH, defined as either:

  1. Ongoing PPH and a systolic blood pressure equal to or less than 80 mm Hg, or
  2. Ongoing PPH, a systolic blood pressure equal to or less than 90 mg Hg and the administration of vasoactive drugs, or
  3. Ongoing PPH and a systolic blood pressure equal to or less than 90 mg Hg as well as a pulse greater than or equal to 120 beats per minute recorded simultaneously

and

* Consent, Deferred consent since 3rd September 2024

Exclusion Criteria:

* Prior cardiac arrest
* Intra-abdominal pregnancy

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse outcome | 42 days
  The proportion of participants with a composite outcome of either maternal death (=death within 42 days post-partum) or emergency hysterectomy

SECONDARY OUTCOMES:
Adverse outcome excluding 'inevitable' hysterectomies | 42 days
  The proportion of participants with a composite outcome of either maternal death (=death within 42 days post-partum) or emergency hysterectomy due to either an irreparable uterine rupture, a pathological placenta growing into the uterus (placenta accreta, increta or percreta) or a pathological uterus, such as a bicorne uterus or one with very large fibroids
Number of AEs and SAEs | 42 days
  Safety of REBOA assessed by AEs and SAEs
Maternal death | 42 days
  The proportion of participants with a maternal death
Emergency hysterectomy | 42 days
  The proportion of participants with emergency hysterectomy
Acute kidney injury | 42 days
  The proportion of participants with acute kidney injury
Transfusions | 42 days
  The number of blood transfusion units
Hemoglobin | 42 days
  Post-partum hemoglobin concentration at day 0, 3 and 42

OTHER OUTCOMES:
REBOA insertion time | 1 day
  Time to insert the REBOA

CONTACTS AND LOCATIONS:
Overall Officials: Thorkild Tylleskar, MD, PhD, Principal Investigator — University of Bergen, Norway
Locations (1):
- Kawempe National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stensaeth KH, Sovik E, Haig IN, Skomedal E, Jorgensen A. Fluoroscopy-free Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) for controlling life threatening postpartum hemorrhage. PLoS One. 2017 Mar 29;12(3):e0174520. doi: 10.1371/journal.pone.0174520. eCollection 2017. PMID 28355242
- [Background] Webster LA, Little O, Villalobos A, Nguyen J, Nezami N, Lilly M, Dariushnia S, Gandhi R, Kokabi N. REBOA: Expanding Applications From Traumatic Hemorrhage to Obstetrics and Cardiopulmonary Resuscitation, From the AJR Special Series on Emergency Radiology. AJR Am J Roentgenol. 2023 Jan;220(1):16-22. doi: 10.2214/AJR.22.27932. Epub 2022 Aug 3. PMID 35920708
- [Background] Brede JR, Sovik E, Rehn M. Resuscitative endovascular balloon occlusion of the aorta: the postpartum haemorrhage perspective. Crit Care. 2022 Mar 11;26(1):57. doi: 10.1186/s13054-022-03942-0. No abstract available. PMID 35277189
- [Background] Brede JR, Rehn M. The end of balloons? Our take on the UK-REBOA trial. Scand J Trauma Resusc Emerg Med. 2023 Oct 31;31(1):69. doi: 10.1186/s13049-023-01142-5. PMID 37908007